CLINICAL TRIAL: NCT02870504
Title: Clinical Study of Laser Peripheral Iridoplasty on Different Sites of Iris
Brief Title: Clinical Study of LPI on Different Sites of Iris
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Maosong Xie, Principal Investigator, First Affiliated Hospital of Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: [2016]102-1
Record Dates: First submitted 2016-08-10; First posted 2016-08-17 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Glaucoma
Keywords: laser peripheral iridoplasty; treatment
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- corneoscleral limbus group (Experimental): Laser spot locates on the corneoscleral limbus.
  Interventions: Procedure: Corneoscleral limbus group
- One spot group (Experimental): Laser spot locates on one spot away from the corneoscleral limbus
  Interventions: Procedure: one spot group
- Two spots group (Experimental): Laser spot locates on two spots away from the corneoscleral limbus
  Interventions: Procedure: two spots group

INTERVENTIONS:
Procedure: Corneoscleral limbus group — Laser spot locates on the corneoscleral limbus
  Arms: corneoscleral limbus group
Procedure: one spot group — Laser spot locates on one spot away from the corneoscleral limbus
  Arms: One spot group
Procedure: two spots group — Laser spot locates on two spots away from the corneoscleral limbus
  Arms: Two spots group

SUMMARY:
Glaucoma is the second cause of blindness worldwide. Laser peripheral iridoplasty (LPI) is a simple and effective treatment for angle closure glaucoma. LPI can widen or reopen an existing angle close or angle adhesion in order to reduce the risk of attack of the angle closure glaucoma. However, there are very little research on the laser site, laser wavelengths, laser energy and laser spot intervals. The purpose of this study is to determine the optimum laser site of LPI.

DETAILED DESCRIPTION:
Glaucoma is the second cause of blindness worldwide. Laser peripheral iridoplasty (LPI) is a simple and effective treatment for angle closure glaucoma. LPI can widen or reopen an existing angle close or angle adhesion in order to reduce the risk of attack of the angle closure glaucoma. However, there are very little research on the laser site, laser wavelengths, laser energy and laser spot intervals.

The purpose of this study is to determine the optimum laser site of LPI. Before and 7days, 1 month, 3 months after LPI, the structure of anterior chamber, including angle anterior chamber depth(ACD), angle of anterior chamber (AA), anterior chamber angle opening distance 750(AOD750) are measured with ultrasound biomicroscopy. Before and 7days, 1 month, 3 months after LPI, the outflow resistance of aqueous humor are evaluated with C value. Before and 1hour, 1days, 3day, 7days, 1 month, 3 months after LPI, intraocular pressure are measured with Goldmann tonometry. Before and 3 months after LPI, retinal nerve layer thickness and the optic disc cup disc ratio are measure with optical coherence tomography.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary angle closure suspect (PACS), primary angle closure (PAC) or primary angle closure glaucoma (PACG).
* PACS is diagnosed in eyes with an occludable angle but no other abnormality.
* PAC is diagnosed in eyes with an occludable angle, normal optic discs and visual fields and any of the following: raised IOP (>19 mm Hg), PAS, pigment smearing in the superior angle, or sequelae of acute angle closure (iris whirling or glaucomatous fleck).
* PACG is diagnosed in eyes with an occludable angle and glaucomatous optic neuropathy. Evidence of glaucomatous optic neuropathy is defined as a cup: disc ratio (CDR) of >0.7 or >0.2 CDR asymmetry.
* An occludable angle is defined as one in which three quarters of the posterior pigmented trabecular meshwork is not visible on viewing with a Goldmann two mirror lens in the primary position of gaze without indentation.

Exclusion Criteria:

* Patients with previous ocular surgery, and those with secondary angle closure, such as lens intumescence or subluxation, iris neovascularisation and a history of uveitis.
* Patients who have systemic contraindications to medical therapy (including renal impairment, sulfur allergy, asthma and heart failure), pre-existing corneal opacities obstructing laser access to more than one quadrant of the peripheral iris and single-eyed patients are also excluded.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change of anterior chamber angle(AA) | Baseline and 3 months after LPI
  Anterior chamber angle (AA) is measured with ultrasound biomicroscopy.

SECONDARY OUTCOMES:
Change of anterior chamber angle opening distance 750(AOD750) | Baseline and 3 months after LPI
  Anterior chamber angle opening distance 750(AOD750) is measured with ultrasound biomicroscopy.
Change of anterior chamber depth(ACD) | Baseline and 3 months after LPI.
  Anterior chamber depth(ACD) is measured with ultrasound biomicroscopy.
Change of intraocular pressure (IOP) | Baseline and 1hour, 1days, 3day, 7days, 1 month, 3 months after LPI.
  IOP is measured with Goldmann tonometry.
Change of C value | Baseline and 7days, 1 month, 3 months after LPI.
  IOP is measured with Schφtz tonometry.
Change of retinal nerve layer thickness | Baseline and 3 months after LPI.
  Retinal nerve layer thickness is measured with optical coherence tomography.
Change of optic disc cup disc ratio | Baseline and 3 months after LPI.
  Optic disc cup disc ratio is measured with optical coherence tomography.
Change of mean defect | Baseline and 3 months after LPI.
  Mean defect is measured with computer perimetry.
Change of mean sensitivity | Baseline and 3 months after LPI.
  Mean sensitivity is measured with computer perimetry.
Change of scotoma | Baseline and 3 months after LPI.
  Scotoma is measured with computer perimetry.

CONTACTS AND LOCATIONS:
Overall Officials: Maosong Xie, doctor, Study Chair — Department of ophthalmology, First Affilited Hospital of Fujian Medical University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lai J, Choy BN, Shum JW. Management of Primary Angle-Closure Glaucoma. Asia Pac J Ophthalmol (Phila). 2016 Jan-Feb;5(1):59-62. doi: 10.1097/APO.0000000000000180. PMID 26886121
- [Background] Narayanaswamy A, Baskaran M, Perera SA, Nongpiur ME, Htoon HM, Tun TA, Wong TT, Goh D, Su DH, Chew PT, Ho CL, Aung T. Argon Laser Peripheral Iridoplasty for Primary Angle-Closure Glaucoma: A Randomized Controlled Trial. Ophthalmology. 2016 Mar;123(3):514-21. doi: 10.1016/j.ophtha.2015.11.002. Epub 2015 Dec 23. PMID 26707418
- [Background] Marchini G, Chemello F, Berzaghi D, Zampieri A. New findings in the diagnosis and treatment of primary angle-closure glaucoma. Prog Brain Res. 2015;221:191-212. doi: 10.1016/bs.pbr.2015.05.001. Epub 2015 Jun 30. PMID 26518079
- [Background] Sng CC, Aquino MC, Liao J, Zheng C, Ang M, Chew PT. Anterior segment morphology after acute primary angle closure treatment: a randomised study comparing iridoplasty and medical therapy. Br J Ophthalmol. 2016 Apr;100(4):542-8. doi: 10.1136/bjophthalmol-2015-307087. Epub 2015 Aug 20. PMID 26294102
- [Background] Wright C, Tawfik MA, Waisbourd M, Katz LJ. Primary angle-closure glaucoma: an update. Acta Ophthalmol. 2016 May;94(3):217-25. doi: 10.1111/aos.12784. Epub 2015 Jun 27. PMID 26119516
- [Background] Fu J, Qing GP, Wang NL, Wang HZ. Efficacy of laser peripheral iridoplasty and iridotomy on medically refractory patients with acute primary angle closure: a three year outcome. Chin Med J (Engl). 2013 Jan;126(1):41-5. PMID 23286475
- [Background] Lee JR, Choi JY, Kim YD, Choi J. Laser peripheral iridotomy with iridoplasty in primary angle closure suspect: anterior chamber analysis by pentacam. Korean J Ophthalmol. 2011 Aug;25(4):252-6. doi: 10.3341/kjo.2011.25.4.252. Epub 2011 Jul 22. PMID 21860572
- [Background] Mochizuki H, Takenaka J, Sugimoto Y, Takamatsu M, Kiuchi Y. Comparison of the prevalence of plateau iris configurations between angle-closure glaucoma and open-angle glaucoma using ultrasound biomicroscopy. J Glaucoma. 2011 Jun-Jul;20(5):315-8. doi: 10.1097/IJG.0b013e3181e3d2da. PMID 20577108